CLINICAL TRIAL: NCT03142191
Title: A Phase 2, 24-Week, Randomized, Double-blind, Placebo-controlled, Multicenter Study, With an 80-Week Active Treatment Extension, to Evaluate the Efficacy and Safety of CC-90001 in Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: A Study to Evaluate the Efficacy and Safety of CC-90001 in Subjects With Idiopathic Pulmonary Fibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-90001-IPF-001; 2016-003473-17 (EudraCT Number); U1111-1192-8549 (Registry Identifier: WHO)
Record Dates: First submitted 2017-04-24; First posted 2017-05-05 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Idiopathic Pulmonary Fibrosis; Fibrosis; Idiopathic Interstitial Pneumonias; Pathologic Processes; Lung Diseases, Interstitial; Lung Diseases; Respiratory Tract Diseases
Keywords: Idiopathic Pulmonary Fibrosis (IPF); Pulmonary Fibrosis; CC-90001; Safety; Efficacy; IPF; idiopathic pulmonary fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Fibrosis; Idiopathic Interstitial Pneumonias; Pathologic Processes; Lung Diseases, Interstitial; Lung Diseases; Respiratory Tract Diseases; Pulmonary Fibrosis | interventions — CC-90001

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CC-90001 400 mg PO QD (Experimental): 55 subjects will be randomized to CC-90001 400mg
  Interventions: Drug: CC-90001
- CC-90001 200 mg PO QD (Experimental): 55 subjects will be randomized to CC-90001 200mg
  Interventions: Drug: CC-90001
- Placebo PO QD (Placebo Comparator): 55 subjects will be randomized to placebo
  Interventions: Other: Placebo
- CC-90001 400 mg PO QD- Sub-Study (Experimental): 30 subjects will be randomized to CC-90001 400mg
  Interventions: Drug: CC-90001
- Placebo PO QD- Sub-Study (Placebo Comparator): 15 subjects will be randomized to placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CC-90001 — CC-90001 is a potent, selective inhibitor of JNK.
  Arms: CC-90001 200 mg PO QD; CC-90001 400 mg PO QD; CC-90001 400 mg PO QD- Sub-Study
Other: Placebo — Placebo
  Arms: Placebo PO QD; Placebo PO QD- Sub-Study

SUMMARY:
This is a Phase 2, multicenter, multinational, randomized, double-blind, placebo-controlled study evaluating the efficacy, safety, pharmacokinetics (PK), quality of life and exploratory pharmacodynamics (PD) of two treatment doses of CC-90001, 200 mg and 400 mg, compared with placebo, when delivered once daily per os (PO) in subjects with idiopathic pulmonary fibrosis (IPF). This study is designed to assess response to treatment by using measures of lung function, disease progression, fibrosis on radiography, and patient-reported outcomes. It will also assess dose response.

DETAILED DESCRIPTION:
Approximately 165 adult male and female subjects with a confirmed diagnosis of Idiopathic pulmonary fibrosis (IPF) (according to the most recent IPF guideline for diagnosis and management) will be randomized 1:1:1 (55 subjects per arm) to treatment with oral CC-90001or matching placebo for an initial 24 weeks.

The randomization will be stratified based on the concurrent administration of SOC (Yes/No). Subjects completing the 24-week Double-blind Treatment Phase will continue onto the 80-week Active Treatment Extension Phase. At Week 24, all subjects originally randomized to receive placebo will be re-randomized 1:1 to blinded CC-90001 (200 mg or 400 mg PO QD). During the 80-week Active Treatment Extension Phase, all subjects not on concurrent SOC therapy will have the opportunity, if deemed appropriate by the Investigator, to receive allowed standard of care (SOC).

The exploratory Progressive Pulmonary Fibrosis (PPF) sub study will evaluate the efficacy, safety, PK, quality of life and exploratory PD of one PO treatment dose regimen of CC-90001, compared with placebo, for an initial 24 weeks of treatment, in subjects with PPF and long-term safety in the 80-week Active Treatment Extension Phase when all PPF subjects will receive CC-90001. Approximately 45 non-SOC subjects will be randomized in this sub study.

All subjects who complete the study treatment phases and those subjects who discontinue investigational product (IP) prior to the completion of the study will participate in the 4-week Post-treatment Observational Follow-up Phase.

The study will be conducted in compliance with the International Council Harmonisation (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use/Good Clinical Practice (GCP) and applicable regulatory requirements.

An external DMC, comprised of independent physician experts and a statistician who are not affiliated with the Sponsor and for whom there is no identified conflict of interest will be responsible for safeguarding study participants' interests and for monitoring the overall conduct of the study.

ELIGIBILITY:
Inclusion Criteria:

Subject understands and has voluntarily signed and dated an informed consent form

1. Subject is male or female ≥ 40 years of age
2. Diagnosis of IPF is supported by HRCT and historical lung biopsy (surgical lung biopsy [SLB] or cryobiopsy) if available according to guidelines.
3. No features supporting an alternative diagnosis on transbronchial biopsy, bronchoalveolar lavage (BAL), or SLB, if performed.
4. Percent predicted forced vital capacity (% FVC) ≥ 45% and ≤ 95% at Screening
5. Percent predicted diffusion capacity of the lung for carbon monoxide (DLCO) ≥ 25% and ≤ 90% predicted at Screening.
6. Able to walk ≥ 150 meters during the 6-minute walk test (6MWT) at Screening
7. Females of childbearing potential (FCBP) must commit to true abstinence or agree to use two effective birth control methods.
8. Male subjects must practice true abstinence or use a barrier method of contraception.
9. Additional inclusion criteria apply.

Progressive Pulmonary Fibrosis (PPF) Sub-Study:

1. Met all inclusion criteria described for IPF subjects other than Inclusion Criterion 5.
2. Features of diffuse fibrosing lung disease of > 10% on HRCT by central reading.
3. Investigator-documented ≥ 5% annualized relative decline in FVC in past 24 months from Screening Visit 1

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject with a QTcF > 450 msec.
3. Evidence of clinically relevant airways obstruction at Screening.
4. Subjects using therapy targeted to treat IPF.
5. History of latent or active TB, unless there is medical record documentation of successful completion of a standard course of treatment
6. History of hepatitis B and/or hepatitis C, including those considered successfully treated/cured
7. Pregnancy or lactation.
8. Additional exclusion criteria apply.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2017-07-26 (Actual); Primary Completion 2021-12-24 (Actual); Study Completion 2021-12-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (112):
- United States (21):
  - Loma Linda Univ Medical Center, Loma Linda, California
  - Cedars Sinai Medical Center Rheumatology, Los Angeles, California
  - Local Institution - 514, Sacramento, California
  - University of California Davis Health System, Sacramento, California
  - Stanford University Pulmonary and Critical Care Clinic, Stanford, California
  - University of Florida, Gainesville, Florida
  - University of Miami and Sylvester Cancer Center, Miami, Florida
  - University of Louisville, Louisville, Kentucky
  - The Lung and Research Center, LLC, Chesterfield, Missouri
  - Mt. Sinai School of Medicine, New York, New York
  - Duke University Health System - Duke Pulmonary Transplant Clinic, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Pulmonary & Sleep Center of Oklahoma, Tulsa, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Local Institution - 502, Dallas, Texas
  - University of Utah Health Care, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont
- Australia (12):
  - Local Institution - 608, Camperdown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Mater Medical Centre, South Brisbane, Queensland
  - Local Institution - 601, Adelaide, South Australia
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Local Institution - 605, Parkville, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Institute for Respiratory Health Inc, Nedlands, Western Australia
  - St Vincent Hospital - Sydney, Darlinghurst
- Brazil (7):
  - Clinica de Pneumologia S/S, Goiânia, Goiás
  - Irmandade da Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital Ernesto Dornelles, Porto Alegre
  - Universidade Federal do Rio de Janeiro (UFRJ)-Hospital Universitario Clementino Fraga Filho (HUCFF), Rio de Janeiro
  - Faculdade de Medicina do ABC, Santo André
  - Incor - Instituto do Coracao HCFMUSP, São Paulo
- Canada (6):
  - Kelowna & Respiratory Allergy Clinic, Kelowna, British Columbia
  - Local Institution - 621, Kelowna, British Columbia
  - Local Institution - 620, Vancouver, British Columbia
  - The Lung Centre Respiratory Clinic - Vancouver General Hospital Location, Vancouver, British Columbia
  - Dr. Syed Anees Medicine Professional Corporation, Windsor, Ontario
  - Local Institution - 623, Windsor, Ontario
- Colombia (4):
  - Centro de Reumatologia y Ortopedia SAS, Barranquilla
  - Local Institution - 631, Bogotá
  - Centro Especializado en Enfermedades Pulmonares, Bogotá
  - Centro Medico Imbanaco, Cali
- Germany (6):
  - Helios Klinikum Emil Von Behring, Berlin
  - Ruhrlandklinik University Hospital, Essen
  - AGAPLESION EV. KRANKENHAUS MITTELHESSEN gGmbH, Giessen
  - Local Institution - 642, Giessen
  - Universitatsklinikum Heidelberg, Heidelberg
  - Waldburg-Zeil Kliniken -Fachkliniken Wangen, Wangen
- Greece (5):
  - Democritus University of Thrace, Alexandroupoli
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - University General Hospital Attikon, Haidari
  - University of Crete - University General Hospital of Heraklion, Heraklion
  - General Hospital of Heraklion Benizeleio Pananeio, Heraklion
- Romania (2):
  - Spitalul Clinic de Pneumoftiziologie Leon Daniello Cluj Napoca, Cluj-Napoca
  - Spitalul Clinic de Boli Infectioase si Pneumoftiziologie Dr. Victor Babes Timisoara, Timișoara
- Russia (17):
  - City clinical hospital No 9, Izhevsk
  - Federal State Budgetary Scientific Institution Research Institute for Complex Issues of Cardiovascul, Kemerovo
  - TSBIH Territorial Clinical Hospital, Krasnoyarsk
  - Russian Academy of Medical Sciences RAMS - Central Scientific Research Institute of Tuberculosis CTR, Moscow
  - Federal Medico-Biological Agency FMBA - Federal Research Clinical Center FGUZ Clinical Hospital No., Moscow
  - Local Institution - 666, Nizhny Novgorod
  - Nizhny Novgorod Research Institute of Hygiene and Occupational Pathology, Nizhny Novgorod
  - Republican Hospital, Petrozavodsk
  - FSBHI Clincial Research Institute of Phithisioplulmonoloyg, Saint Petersburg
  - Local Institution - 667, Saint Petersburg
  - Vvedenskaya Hospital, Saint Petersburg
  - Saint-Petersburg State Institution of Healthcare, Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Local Institution - 675, Saratov
  - Saratov Regional Clinical Hospital, Saratov
  - SAIH of Yaroslavl region Clinical Hospital for Emergency Medical Care n.a. N.V.Solovyev, Yaroslavl
  - Ural State Medical Academy - Medical Association Novaya Bolnitsa, Yekaterinburg
- Taiwan (4):
  - Buddhist Dalin Tzu Chi General Hospital, Dalin
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei, Zhongzheng Dist.
- Turkey (Türkiye) (5):
  - Ege Universitesi Tip Fakultesi Hastanesi Ege University Medical Faculty Hospital, Bornova
  - Local Institution - 681, Bornova
  - Uludag Universitesi Tip Fakultesi, Bursa
  - Istanbul Universitesi - Cerrahpasa Tip Fakultesi Cerrahpasa Medical Faculty, Istanbul
  - Izmir Dr.Suat Seren Chest Diseases Hospital, Izmir
- Ukraine (6):
  - Communal Institution Dnipropetrovsk City Clinical Hospital #6 of Dnipropetrovsk Regional Council, Dnipro
  - Regional Phthisiopulmonological Center, Ivano-Frankivsk
  - Kharkiv City Clinical Hospital #13, Kharkiv
  - CI of Healthcare RCH - Center of Medical Emergency and Accident Medicine, Kharkiv
  - State Institution National Scientific Center of Radiation Medicine of NAMS of Ukraine, Kyiv
  - SI F.H.Yanovskyi National Institute of Phthisiatry and Pulmonology of Academy of Medical Sciences, Kyiv
- United Kingdom (17):
  - Birmingham Chest Clinic, Birmingham
  - Hull and East Yorkshire Hospitals NHS Trust - Castle Hill Hospital, Cottingham
  - Hinchingbrooke Hospital, Huntingdon
  - The Leeds Teaching Hospitals NHS Trust - St James's University Hospital, Leeds
  - University Hospitals of Leicester NHS Trust - Glenfield Hospital - Institute for Lung Health ILH, Leicester
  - Aintree University Hospital, Liverpool (Walton Centre)
  - University Hospital Llandough, Llandough
  - University College London Hospitals, London
  - Local Institution - 598, Newcastle
  - Royal Victoria Infirmary, Newcastle
  - Local Institution - 697, Norwich
  - Norfolk and Norwich University Hospital, Norwich
  - The University of Nottingham - Nottingham Respiratory Research Unit NRRU, Nottingham
  - Salford Royal, Salford
  - Southampton General Hospital, Southhampton
  - Local Institution - 694, Westbury-on-Trym/ Bristol
  - Southmead Hospital, Westbury-on-Trym/ Bristol

REFERENCES:
- [Derived] Mattos WLLD, Khalil N, Spencer LG, Bonella F, Folz RJ, Rolf JD, Mogulkoc N, Lancaster LH, Jenkins RG, Lynch DA, Noble PW, Maher TM, Cottin V, Senger S, Horan GS, Greenberg S, Popmihajlov Z. Phase 2, Double-Blind, Placebo-controlled Trial of a c-Jun N-Terminal Kinase Inhibitor in Idiopathic Pulmonary Fibrosis. Am J Respir Crit Care Med. 2024 Aug 15;210(4):435-443. doi: 10.1164/rccm.202310-1907OC. PMID 38484130
- [Derived] Popmihajlov Z, Sutherland DJ, Horan GS, Ghosh A, Lynch DA, Noble PW, Richeldi L, Reiss TF, Greenberg S. CC-90001, a c-Jun N-terminal kinase (JNK) inhibitor, in patients with pulmonary fibrosis: design of a phase 2, randomised, placebo-controlled trial. BMJ Open Respir Res. 2022 Jan;9(1):e001060. doi: 10.1136/bmjresp-2021-001060. PMID 35058236
- [Derived] Nagy MA, Hilgraf R, Mortensen DS, Elsner J, Norris S, Tikhe J, Yoon W, Paisner D, Delgado M, Erdman P, Haelewyn J, Khambatta G, Xu L, Romanow WJ, Condroski K, Bahmanyar S, McCarrick M, Benish B, Blease K, LeBrun L, Moghaddam MF, Apuy J, Canan SS, Bennett BL, Satoh Y. Discovery of the c-Jun N-Terminal Kinase Inhibitor CC-90001. J Med Chem. 2021 Dec 23;64(24):18193-18208. doi: 10.1021/acs.jmedchem.1c01716. Epub 2021 Dec 13. PMID 34894681
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants in the placebo arm during treatment period were re-randomized during the active treatment period to receive either CC-90001 200mg or CC-90001 400mg.
  1 participant in the active treatment period did not have the end of study form filled out and therefore was listed in the missing row.
Groups:
- CC-90001 200mg (IPF Study): CC-90001 200mg PO QD
- CC-90001 400mg (IPF Study); CC-90001 400mg (PPF Sub-Study): CC-90001 400mg PO QD
- Placebo (IPF Study); Placebo (PPF Sub-Study): Placebo
Period: Placebo Controlled Period
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo (IPF Study) | CC-90001 400mg (PPF Sub-Study) | Placebo (PPF Sub-Study)
Started | 39 | 37 | 36 | 15 | 8
Completed | 32 | 28 | 31 | 15 | 7
Not Completed | 7 | 9 | 5 | 0 | 1
Not completed — Death | 0 | 1 | 1 | 0 | 0
Not completed — Adverse Event | 4 | 5 | 1 | 0 | 0
Not completed — Progressive Disease | 1 | 0 | 1 | 0 | 0
Not completed — Withdrawal by participant | 1 | 3 | 2 | 0 | 1
Not completed — Other Reasons | 1 | 0 | 0 | 0 | 0
Period: Active Treatment Extension Period
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo (IPF Study) | CC-90001 400mg (PPF Sub-Study) | Placebo (PPF Sub-Study)
Started | 31 | 27 | 30 | 15 | 6
CC-90001 200mg (Participants who were in the placebo arm during treatment period and are now taking CC-90001 200mg) | 0 | 0 | 15 | 0 | 3
CC-90001 400mg (Participants who were in the placebo arm during treatment period and are now taking CC-90001 400mg) | 0 | 0 | 15 | 0 | 3
Completed | 5 | 13 | 15 | 3 | 0
Not Completed | 26 | 14 | 15 | 12 | 6
Not completed — Death | 2 | 1 | 1 | 1 | 0
Not completed — Adverse Event | 6 | 5 | 4 | 1 | 0
Not completed — Progressive Disease | 10 | 5 | 4 | 1 | 2
Not completed — Withdrawal by participant | 2 | 0 | 3 | 1 | 1
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 0
Not completed — Other Reasons | 3 | 3 | 3 | 8 | 3
Not completed — Unknown, participant missing | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo (IPF Study) | CC-90001 400mg (PPF Sub-Study) | Placebo (PPF Sub-Study) | Total
Number analyzed (Participants) | 39 | 37 | 36 | 15 | 8 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 7 | 5 | 8 | 5 | 36
  >=65 years | 28 | 30 | 31 | 7 | 3 | 99
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 6 | 6 | 4 | 35
  Male | 28 | 29 | 30 | 9 | 4 | 100
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 3 | 0 | 0 | 11
  Not Hispanic or Latino | 35 | 33 | 32 | 15 | 8 | 123
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 38 | 35 | 35 | 15 | 8 | 131
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage Point Difference in % Predicted Forced Vital Capacity (FVC).
Description: Mean change from baseline in percentage point difference in % predicted forced vital capacity (FVC)
  FAS population is defined as all randomized participants who received at least one dose of the investigational product.
  Baseline is defined as day 1 of treatment.
Time Frame: from baseline to week 24
Population: Full Analysis Set in IPF Cohort
Measure: Mean (Standard Deviation); unit: Percentage Point
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo (IPF Study)
Number analyzed (Participants) | 39 | 37 | 36
Percentage Point
  Week 1: number analyzed (Participants) | 38 | 32 | 36
  Week 1 | 0.5 (3.04) | 0.6 (2.87) | -0.9 (3.51)
  Week 4: number analyzed (Participants) | 38 | 34 | 34
  Week 4 | 0.3 (4.65) | 1.7 (3.90) | -1.4 (3.75)
  Week 8: number analyzed (Participants) | 35 | 30 | 34
  Week 8 | 0.5 (5.70) | 2.4 (3.98) | -1.7 (3.75)
  Week 12: number analyzed (Participants) | 36 | 28 | 35
  Week 12 | -0.6 (4.83) | 2.0 (3.70) | -2.5 (4.57)
  Week 16: number analyzed (Participants) | 33 | 28 | 33
  Week 16 | -1.7 (5.55) | 1.0 (5.27) | -2.0 (4.43)
  Week 20: number analyzed (Participants) | 33 | 29 | 31
  Week 20 | -1.2 (3.92) | 0.6 (4.55) | -2.7 (6.60)
  Week 24: number analyzed (Participants) | 32 | 29 | 30
  Week 24 | -2.3 (4.96) | -0.5 (4.77) | -2.5 (4.85)

2. Secondary Outcome: Mean Change From Baseline in Absolute Forced Vital Capacity (FVC).
Description: Mean change from baseline in absolute FVC in the full analysis set (FAS) population.
  FAS population is defined as all randomized participants who received at least one dose of the investigational product.
  Baseline is defined as day 1 of treatment.
Time Frame: from baseline to week 24
Population: Full Analysis Set participants with evaluable measures in IPF cohort at week 24
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo (IPF Study)
Number analyzed (Participants) | 32 | 29 | 30
mL | -74.9 (162.58) | -6.8 (170.39) | -88.3 (176.80)

3. Secondary Outcome: Mean Change in Distance Walked in the 6-minute Walk Test (6MWT)
Description: Mean change in distance walked in the 6-minute Walk Test (6MWT)
  The 6MWT measures the distance a participant is able to walk on a hard, flat surface, over a total of six minutes.
  The time points which will be measured are from baseline to Week 24, Extension Week 52, Extension Week 76, Extension Week 104, Week 24 to extension (Ext) Week 52 and Week 24 to Ext Week 104
  FAS population is defined as all randomized participants who received at least one dose of the investigational product.
  Baseline is defined as day 1 of treatment. Week 24 is the start of baseline of the active treatment extension period.
Time Frame: From baseline up to week 104
Population: Full Analysis Set in the IPF cohort
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Placebo/CC-90001 200mg (IPF Study): Participants who received placebo in the placebo treatment phase and then CC-90001 200mg PO QD in the active treatment extension phase
- Placebo/CC-90001 400mg (IPF Study): Participants who received placebo in the placebo treatment phase and then CC-90001 400mg PO QD in the active treatment extension phase
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo (IPF Study) | Placebo/CC-90001 200mg (IPF Study) | Placebo/CC-90001 400mg (IPF Study)
Number analyzed (Participants) | 39 | 37 | 36 | 15 | 15
meters
  Week 24: number analyzed (Participants) | 31 | 28 | 29 | 0 | 0
  Week 24 | 6.9 (73.42) | -21.1 (45.80) | -8.1 (49.89) |  |
  Extension Week 52: number analyzed (Participants) | 19 | 16 | 0 | 8 | 11
  Extension Week 52 | -21.9 (82.57) | -15.9 (46.42) |  | -30.0 (56.69) | -29.1 (94.95)
  Extension Week 76: number analyzed (Participants) | 10 | 10 | 0 | 5 | 6
  Extension Week 76 | -9.7 (58.90) | 3.7 (46.31) |  | 14.4 (25.00) | -42.7 (92.46)
  Extension Week 104: number analyzed (Participants) | 3 | 6 | 0 | 6 | 6
  Extension Week 104 | -15.3 (95.13) | -25.4 (58.73) |  | -18.6 (56.24) | -38.7 (87.80)
  Week 24 to Ext Week 52: number analyzed (Participants) | 18 | 16 | 0 | 8 | 11
  Week 24 to Ext Week 52 | 0.2 (1.02) | 0.7 (1.25) |  | -0.9 (0.88) | 0.7 (1.59)
  Week 24 to Ext Week 104: number analyzed (Participants) | 3 | 6 | 0 | 6 | 6
  Week 24 to Ext Week 104 | 0.0 (1.00) | -0.3 (0.42) |  | 0.6 (1.24) | -0.1 (1.66)

4. Secondary Outcome: Mean Change From Baseline in Dyspnea Rating on Borg Scale
Description: Mean change from baseline in dyspnea rating on Borg Scale after the 6MWT.
  The Borg scale ranges from 0 to 10. Where 0 is no dyspnea and a 10 is extremely strong dyspnea. The lower the number the better.
  The time points which will be measured are from baseline to Week 24, Extension Week 52, Extension Week 76, Extension Week 104, Week 24 to extension (Ext) Week 52 and Week 24 to Ext Week 104
  FAS population is defined as all randomized participants who received at least one dose of the investigational product.
  Baseline is defined as day 1 of treatment. Week 24 is the start of baseline of the active treatment extension period.
Time Frame: From baseline up to week 104
Population: Full Analysis Set in the IPF cohort
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo (IPF Study) | Placebo/CC-90001 200mg (IPF Study) | Placebo/CC-90001 400mg (IPF Study)
Number analyzed (Participants) | 39 | 37 | 36 | 15 | 15
Score on a Scale
  Week 24: number analyzed (Participants) | 31 | 27 | 29 | 0 | 0
  Week 24 | 0.4 (1.38) | 0.1 (1.39) | 0.0 (1.55) |  |
  Extension Week 52: number analyzed (Participants) | 18 | 16 | 0 | 8 | 11
  Extension Week 52 | 0.9 (1.32) | 1.3 (1.48) |  | 0.1 (0.68) | 1.0 (1.93)
  Extension Week 76: number analyzed (Participants) | 10 | 10 | 0 | 5 | 6
  Extension Week 76 | -0.2 (1.53) | 1.2 (1.30) |  | -0.7 (1.30) | -0.5 (1.52)
  Extension Week 104: number analyzed (Participants) | 3 | 6 | 0 | 6 | 6
  Extension Week 104 | 1.0 (3.50) | 0.6 (1.15) |  | 1.3 (0.88) | -0.5 (1.52)
  Week 24 to Ext Week 52: number analyzed (Participants) | 18 | 16 | 0 | 8 | 11
  Week 24 to Ext Week 52 | 0.7 (1.71) | 1.1 (1.53) |  | -0.1 (0.64) | 1.5 (2.25)
  Week 24 to Ext Week 104: number analyzed (Participants) | 3 | 6 | 0 | 6 | 6
  Week 24 to Ext Week 104 | 1.8 (2.57) | -0.1 (1.02) |  | 0.3 (0.52) | 0.2 (2.25)

5. Secondary Outcome: Percentage of Participants Who Had Disease Progression
Description: Disease progression is defined as one or more of the following:
  * Death from respiratory failure,
  * Absolute decrease of ≥ 10% from baseline in % predicted FVC at two consecutive evaluations at a minimum of 4 weeks between evaluations
  * Decrease from baseline of ≥ 50 meters in 6MWT distance (in the absence of a readily explainable cause, such as injury or trauma).
  * Unexplained worsening hypoxemia (an absolute decrease from baseline of 4% or more in arterial oxygen saturation by pulse oximetry [SpO2]).
  FAS population is defined as all randomized participants who received at least one dose of the investigational product.
  Baseline is defined as day 1 of treatment.
Time Frame: From Baseline up to week 24
Population: Full analysis set in IPF Cohort
Measure: Number; unit: Percentage of participants
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo (IPF Study)
Number analyzed (Participants) | 39 | 37 | 36
Percentage of participants | 23.1 | 27.0 | 25.0

6. Secondary Outcome: Mean Change From Baseline in Total Score and Domains on the Saint George's Respiratory Questionnaire (SGRQ)
Description: The SGRQ is a quality of life health questionnaire that has been validated in IPF. It consists of 76 items in three domains:
  * Symptoms
  * Activity
  * Impact of disease on daily life
  A total score is calculated from 0 (no health impairment) to 100 (maximum health impairment). In addition to the total score, there is also a score for each domain: symptoms, activity, and impact which are scored 0-100. Each component score is derived by dividing the summed weights, unique for all questions, by the maximum possible weight.
Time Frame: From Baseline up to week 24
Population: Full analysis set with evaluable SGRQ measures in IPF Cohort
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo (IPF Study)
Number analyzed (Participants) | 28 | 23 | 27
Score on a Scale
  Activity | 2.1 (16.95) | -6.5 (12.72) | -4.5 (13.04)
  Impact of disease on daily life | -1.9 (19.31) | -8.6 (19.17) | -1.2 (20.59)
  Symptoms | 2.0 (21.10) | -11.8 (17.57) | -8.3 (20.63)
  Total | -0.3 (16.84) | -8.6 (15.44) | -3.7 (15.99)

7. Secondary Outcome: Mean Change From Baseline in The University of California San Diego Shortness of Breath Questionnaire (UCSD-SOBQ)
Description: The UCSD-SOBQ is a 24-item dyspnea questionnaire that asks participants to rate themselves from 0 ("Not at all") to 5 ("Maximally or unable to do because of breathlessness") in two areas: 1) how short of breath they are while performing various activities (21 items); and 2) how much shortness of breath, fear of hurting themselves by overexerting, and fear of shortness of breath limit them in their daily lives (3 items). If the subject does not routinely perform the activity, they are asked to estimate the degree of shortness of breath anticipated. The UCSD-SOBQ is scored by summing responses across all 24 items to form a total score. Scores range from 0 to 120. The lower the score the better.
Time Frame: From Baseline up to week 24
Population: Full analysis set with evaluable UCSD-SOBQ measures in IPF Cohort
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo (IPF Study)
Number analyzed (Participants) | 26 | 23 | 27
Score on a Scale | 1.1 (17.28) | -3.3 (16.69) | -1.4 (16.19)

8. Secondary Outcome: Number of Participants With Adverse Events at the End of the Active Treatment Phase
Description: Number of participants with Adverse events at the end of the active treatment phase
Time Frame: From re-randomization to end of treatment (approximately 84 weeks)
Population: Re-randomized safety set
Measure: Count of Participants; unit: Participants
Groups:
- Placebo/CC-90001 200mg (PPF Sub-study): Participants who received placebo in the placebo treatment phase and then CC-90001 200mg PO QD in the active treatment extension phase
- Placebo/CC-90001 400mg (PPF Sub-Study): Participants who received placebo in the placebo treatment phase and then CC-90001 400mg PO QD in the active treatment extension phase
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo/CC-90001 200mg (IPF Study) | Placebo/CC-90001 400mg (IPF Study) | CC-90001 400mg (PPF Sub-Study) | Placebo/CC-90001 200mg (PPF Sub-study) | Placebo/CC-90001 400mg (PPF Sub-Study)
Number analyzed (Participants) | 31 | 27 | 15 | 15 | 15 | 3 | 3
Participants
  TEAE | 25 | 23 | 11 | 13 | 11 | 2 | 3
  TEAE related to study treatment | 7 | 13 | 2 | 8 | 1 | 1 | 0
  Serious TEAE | 10 | 6 | 3 | 4 | 2 | 0 | 0
  Serious TEAE related to study Drug | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Severe TEAE | 8 | 7 | 2 | 4 | 2 | 0 | 0
  TEAE leading to Death | 5 | 4 | 2 | 2 | 1 | 0 | 0
  TEA leading to study treatment interruption | 2 | 6 | 1 | 2 | 1 | 0 | 0
  TEAE leading to permanent study treatment discontinuation | 6 | 4 | 0 | 3 | 1 | 0 | 0

9. Secondary Outcome: Number of Participants With Adverse Events in the Placebo Controlled Period
Description: Number of participants with Adverse events
Time Frame: from baseline to re-randomization (approximately 56 weeks for the IPF cohort and 28 weeks for the PPF cohort)
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo (IPF Study) | CC-90001 400mg (PPF Sub-Study) | Placebo (PPF Sub-Study)
Number analyzed (Participants) | 39 | 37 | 36 | 15 | 8
Participants
  TEAE | 30 | 34 | 31 | 8 | 5
  TEAE related to study treatment | 14 | 21 | 14 | 3 | 1
  Serious TEAE | 6 | 4 | 2 | 1 | 0
  Serious TEAE related to study Drug | 1 | 1 | 0 | 0 | 0
  Severe TEAE | 4 | 8 | 3 | 0 | 0
  TEAE leading to Death | 0 | 1 | 2 | 0 | 0
  TEA leading to study treatment interruption | 6 | 3 | 5 | 0 | 2
  TEAE leading to permanent study treatment discontinuation | 5 | 7 | 2 | 0 | 0

10. Secondary Outcome: Number of Participants With Worst Changes in Hematology Laboratory Parameters During the Active Treatment Extension Period
Description: Number of participants with worst changes in hematology laboratory parameters including: basophils, hemoglobin, lymphocytes, neutrophils and platelets.
Time Frame: From re-randomization to end of treatment (approximately 84 weeks)
Population: Re-randomized safety set
Measure: Count of Participants; unit: Participants
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo/CC-90001 200mg (IPF Study) | Placebo/CC-90001 400mg (IPF Study) | CC-90001 400mg (PPF Sub-Study) | Placebo/CC-90001 400mg (PPF Sub-study) | Placebo/CC-90001 200mg (PPF Sub-Study)
Number analyzed (Participants) | 31 | 27 | 15 | 15 | 15 | 3 | 3
Participants
  Basophils - Normal to low: number analyzed (Participants) | 30 | 27 | 14 | 15 | 14 | 3 | 3
  Basophils - Normal to low | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Basophils - Normal to high: number analyzed (Participants) | 30 | 27 | 14 | 15 | 14 | 3 | 3
  Basophils - Normal to high | 5 | 3 | 1 | 1 | 0 | 0 | 0
  Hemoglobin - Normal to low: number analyzed (Participants) | 28 | 24 | 14 | 14 | 14 | 3 | 3
  Hemoglobin - Normal to low | 2 | 2 | 1 | 0 | 1 | 0 | 0
  Hemoglobin - Normal to high: number analyzed (Participants) | 28 | 24 | 14 | 14 | 14 | 3 | 3
  Hemoglobin - Normal to high | 3 | 4 | 2 | 1 | 0 | 0 | 0
  Lymphocytes - Normal to low: number analyzed (Participants) | 28 | 24 | 12 | 14 | 12 | 2 | 3
  Lymphocytes - Normal to low | 2 | 2 | 0 | 1 | 1 | 0 | 0
  Lymphocytes - Normal to high: number analyzed (Participants) | 28 | 24 | 12 | 14 | 12 | 2 | 3
  Lymphocytes - Normal to high | 3 | 5 | 2 | 1 | 0 | 1 | 1
  Neutrophils - Normal to low: number analyzed (Participants) | 28 | 26 | 10 | 12 | 14 | 2 | 2
  Neutrophils - Normal to low | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Neutrophils - Normal to high: number analyzed (Participants) | 28 | 26 | 10 | 12 | 14 | 2 | 2
  Neutrophils - Normal to high | 14 | 11 | 6 | 6 | 1 | 0 | 0
  Platelets - Normal to low: number analyzed (Participants) | 29 | 25 | 13 | 15 | 13 | 3 | 3
  Platelets - Normal to low | 0 | 1 | 0 | 2 | 0 | 0 | 0
  Platelets - Normal to high: number analyzed (Participants) | 29 | 25 | 13 | 15 | 13 | 3 | 3
  Platelets - Normal to high | 0 | 1 | 1 | 0 | 0 | 0 | 0

11. Secondary Outcome: Number of Participants With Worst Changes in Hematology Laboratory Parameters During the in the Placebo Controlled Period
Description: as for outcome 10
Time Frame: from baseline to re-randomization (approximately 56 weeks for the IPF cohort and 28 weeks for the PPF cohort)
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo (IPF Study) | CC-90001 400mg (PPF Sub-Study) | Placebo (PPF Sub-Study)
Number analyzed (Participants) | 39 | 37 | 36 | 15 | 8
Participants
  Basophils - Normal to low: number analyzed (Participants) | 38 | 37 | 36 | 15 | 8
  Basophils - Normal to low | 0 | 0 | 0 | 0 | 0
  Basophils - Normal to high: number analyzed (Participants) | 38 | 37 | 36 | 15 | 8
  Basophils - Normal to high | 3 | 0 | 1 | 3 | 2
  Hemoglobin - Normal to low: number analyzed (Participants) | 36 | 34 | 35 | 15 | 8
  Hemoglobin - Normal to low | 4 | 2 | 1 | 0 | 0
  Hemoglobin - Normal to high: number analyzed (Participants) | 36 | 34 | 35 | 15 | 8
  Hemoglobin - Normal to high | 2 | 2 | 3 | 0 | 0
  Lymphocytes - Normal to low: number analyzed (Participants) | 35 | 34 | 32 | 13 | 7
  Lymphocytes - Normal to low | 1 | 2 | 2 | 3 | 0
  Lymphocytes - Normal to high: number analyzed (Participants) | 35 | 34 | 32 | 13 | 7
  Lymphocytes - Normal to high | 4 | 4 | 2 | 3 | 1
  Neutrophils - Normal to low: number analyzed (Participants) | 34 | 34 | 29 | 14 | 6
  Neutrophils - Normal to low | 1 | 0 | 0 | 1 | 1
  Neutrophils - Normal to high: number analyzed (Participants) | 34 | 34 | 29 | 14 | 6
  Neutrophils - Normal to high | 6 | 10 | 7 | 3 | 2
  Platelets - Normal to low: number analyzed (Participants) | 36 | 34 | 35 | 14 | 8
  Platelets - Normal to low | 0 | 1 | 2 | 0 | 0
  Platelets - Normal to high: number analyzed (Participants) | 36 | 34 | 35 | 14 | 8
  Platelets - Normal to high | 4 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With a Change From Worst Post-baseline in Urinalysis Laboratory Analysis in the Active Treatment Extension Period
Description: Number of participants who had a change from worst post- baseline in urinalysis laboratory analysis for the following measures:
  Erythrocytes, Leukocytes, Tubular Epithelial Cells
Time Frame: From re-randomization to end of treatment (approximately 84 weeks)
Population: Re-Randomized Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo/CC-90001 200mg (IPF Study) | Placebo/CC-90001 400mg (IPF Study) | CC-90001 400mg (PPF Sub-Study) | Placebo/CC-90001 200mg (PPF Sub-Study) | Placebo/CC-90001 400mg (PPF Sub-study)
Number analyzed (Participants) | 31 | 27 | 15 | 15 | 15 | 3 | 3
Participants
  Erythrocytes - Normal to abnormal: number analyzed (Participants) | 4 | 2 | 3 | 2 | 2 | 1 | 1
  Erythrocytes - Normal to abnormal | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Leukocytes - Normal to abnormal: number analyzed (Participants) | 10 | 5 | 5 | 2 | 4 | 0 | 1
  Leukocytes - Normal to abnormal | 2 | 1 | 0 | 0 | 2 | 0 | 1
  Tubular Epithelial Cells - Normal abnormal: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With a Change From Worst Post-baseline in Urinalysis Laboratory Analysis in the Placebo Controlled Period
Description: as for outcome 12
Time Frame: from baseline to re-randomization (approximately 56 weeks for the IPF cohort and 28 weeks for the PPF cohort)
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo (IPF Study) | CC-90001 400mg (PPF Sub-Study) | Placebo (PPF Sub-Study)
Number analyzed (Participants) | 39 | 37 | 36 | 15 | 8
Participants
  Erythrocytes - Normal to Abnormal: number analyzed (Participants) | 7 | 6 | 7 | 4 | 3
  Erythrocytes - Normal to Abnormal | 3 | 0 | 0 | 1 | 0
  Leukocytes - Normal to Abnormal: number analyzed (Participants) | 14 | 12 | 7 | 5 | 2
  Leukocytes - Normal to Abnormal | 4 | 1 | 2 | 2 | 0
  Tubular Epithelial Cells - Normal to Abnormal: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Mean Change From Baseline in Electrocardiogram Measurements in the Active Treatment Extension Period
Description: Mean change from baseline in Electrocardiogram readings for the following measures: QT interval, QTcF interval, QTcB interval, PR interval, QRS duration and RR interval
Time Frame: From re-randomization to 4 week follow up after end of treatment (approximately 84 weeks)
Population: Re-Randomized Safety Set
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo/CC-90001 200mg (IPF Study) | Placebo/CC-90001 400mg (IPF Study) | CC-90001 400mg (PPF Sub-Study) | Placebo/CC-90001 200mg (PPF Sub-study) | Placebo/CC-90001 400mg (PPF Sub-Study)
Number analyzed (Participants) | 31 | 27 | 15 | 15 | 15 | 3 | 3
msec
  QT Interval: number analyzed (Participants) | 16 | 15 | 9 | 8 | 8 | 2 | 2
  QT Interval | -14.3 (29.70) | 0.2 (23.85) | -7.7 (22.23) | -10.9 (22.53) | -3.0 (21.29) | 9.0 (28.28) | 25.0 (26.87)
  QTcF Interval: number analyzed (Participants) | 16 | 15 | 9 | 8 | 8 | 2 | 2
  QTcF Interval | -3.9 (21.13) | 2.2 (18.75) | -3.4 (15.02) | -1.9 (4.94) | 5.6 (26.09) | 14.0 (11.31) | 23.5 (4.95)
  QTcB Interval: number analyzed (Participants) | 16 | 15 | 9 | 8 | 8 | 2 | 2
  QTcB Interval | 1.3 (21.06) | 3.5 (25.53) | -0.7 (19.04) | 2.9 (13.46) | 10.0 (37.36) | 17.5 (31.82) | 22.5 (6.36)
  PR Interval: number analyzed (Participants) | 16 | 14 | 9 | 8 | 7 | 2 | 2
  PR Interval | -9.2 (17.07) | 9.2 (18.63) | -12.8 (6.55) | 3.3 (15.27) | 0.6 (16.27) | 14.5 (28.99) | 2.0 (7.07)
  QRS Duration: number analyzed (Participants) | 16 | 15 | 9 | 8 | 8 | 2 | 2
  QRS Duration | -1.8 (7.11) | 5.1 (14.46) | 1.0 (7.25) | -3.8 (5.60) | 2.1 (7.24) | 2.5 (2.12) | 14.5 (13.44)
  RR Interval: number analyzed (Participants) | 16 | 15 | 9 | 8 | 8 | 2 | 2
  RR Interval | -75.4 (129.46) | -14.0 (148.45) | -25.7 (136.36) | -77.9 (181.66) | -51.4 (167.76) | -28.0 (272.94) | 15.5 (135.06)

15. Secondary Outcome: Mean Change From Baseline in Electrocardiogram Measurements in the Placebo Controlled Period
Description: as for outcome 14
Time Frame: from baseline to week 24
Population: Safety Set
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo (IPF Study) | CC-90001 400mg (PPF Sub-Study) | Placebo (PPF Sub-Study)
Number analyzed (Participants) | 39 | 37 | 36 | 15 | 8
msec
  QT Interval: number analyzed (Participants) | 19 | 19 | 22 | 10 | 2
  QT Interval | -2.9 (22.37) | 0.2 (22.76) | -1.8 (26.23) | -9.6 (30.52) | -15.0 (15.56)
  QTcF Interval: number analyzed (Participants) | 19 | 19 | 22 | 10 | 2
  QTcF Interval | -0.3 (15.12) | -0.9 (13.23) | -2.2 (16.80) | 1.5 (16.83) | 6.0 (1.41)
  QTcB Interval: number analyzed (Participants) | 19 | 19 | 22 | 10 | 2
  QTcB Interval | 0.5 (19.57) | -1.2 (16.57) | -2.4 (18.20) | 7.6 (23.51) | 19.0 (11.31)
  PR Interval: number analyzed (Participants) | 19 | 19 | 22 | 8 | 2
  PR Interval | -5.1 (13.89) | -0.3 (10.84) | -0.8 (12.02) | -5.3 (12.23) | 20.5 (20.51)
  QRS Duration: number analyzed (Participants) | 19 | 19 | 22 | 10 | 2
  QRS Duration | 2.0 (8.86) | 2.1 (9.65) | -0.5 (8.44) | -0.9 (6.74) | -3.0 (4.24)
  RR Interval: number analyzed (Participants) | 20 | 19 | 22 | 10 | 2
  RR Interval | -20.9 (127.25) | 6.5 (127.19) | 13.0 (129.92) | -68.4 (173.55) | -110.5 (78.49)

16. Secondary Outcome: Number of Participants With Worst Increase From Baseline in Blood Pressure in the Active Extension Period
Description: Number of participants with worst increase from baseline in systolic and diastolic blood pressure.
Time Frame: From re-randomization to 4 week follow up after end of treatment (approximately 84 weeks)
Population: Re-Randomized Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo/CC-90001 200mg (IPF Study) | Placebo/CC-90001 400mg (IPF Study) | CC-90001 400mg (PPF Sub-Study) | Placebo/CC-90001 200mg (PPF Sub-study) | Placebo/CC-90001 400mg (PPF Sub-Study)
Number analyzed (Participants) | 31 | 27 | 15 | 15 | 15 | 3 | 3
Participants
  systolic increase from baseline > 10 but ≤ 15 (mild) | 5 | 4 | 3 | 1 | 1 | 0 | 0
  systolic increase from baseline > 15 but ≤ 20 (moderate) | 1 | 4 | 2 | 3 | 0 | 0 | 0
  systolic increase from baseline > 20 (severe) | 4 | 8 | 4 | 4 | 0 | 0 | 1
  diastolic increase from baseline > 5 but ≤ 10 (mild) | 6 | 6 | 7 | 3 | 4 | 1 | 2
  diastolic increase from baseline > 10 but ≤ 15 (moderate) | 5 | 3 | 2 | 4 | 1 | 0 | 0
  diastolic increase from baseline > 15 (severe) | 5 | 6 | 5 | 1 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Worst Increase From Baseline in Blood Pressure in the Placebo-controlled Period
Description: Number of participants with worst increase from baseline in systolic and diastolic blood pressure.
Time Frame: from baseline to re-randomization (approximately 56 weeks for the IPF cohort and 28 weeks for the PPF cohort)
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | CC-90001 200mg (IPF Study) | CC-90001 400mg (IPF Study) | Placebo (IPF Study) | CC-90001 400mg (PPF Sub-Study) | Placebo (PPF Sub-Study)
Number analyzed (Participants) | 39 | 37 | 36 | 0 | 0
Participants
  systolic increase from baseline > 10 but ≤ 15 (mild) | 2 | 0 | 2 |  |
  systolic increase from baseline > 15 but ≤ 20 (moderate) | 3 | 2 | 3 |  |
  systolic increase from baseline > 20 (severe) | 0 | 3 | 0 |  |
  diastolic increase from baseline > 5 but ≤ 10 (mild) | 4 | 2 | 1 |  |
  diastolic increase from baseline > 10 but ≤ 15 (moderate) | 3 | 2 | 1 |  |
  diastolic increase from baseline > 15 (severe) | 2 | 2 | 2 |  |

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: (From first dose to last dose + 28 days): Approximately 84 weeks All-Cause mortality (From randomization to end of study): Approximately 104 weeks
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants.
  The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- CC-90001 200mg IPF Study; Active Treatment Phase CC-90001 200mg Following Placebo IPF Study; Active Treatment Phase CC-90001 200mg Following Placebo PPF Sub-Study: CC-90001 200mg PO QD
- CC-90001 400mg IPF Study; Active Treatment Phase CC-90001 400mg Following Placebo IPF Study; CC-90001 400mg PPF Sub-Study; Active Treatment Phase CC-90001 400mg Following Placebo PPF Sub-Study: CC-90001 400mg PO QD
- Placebo IPF Study; Placebo PPF Sub-Study: Placebo
Arm/Group | CC-90001 200mg IPF Study | CC-90001 400mg IPF Study | Placebo IPF Study | Active Treatment Phase CC-90001 200mg Following Placebo IPF Study | Active Treatment Phase CC-90001 400mg Following Placebo IPF Study | CC-90001 400mg PPF Sub-Study | Placebo PPF Sub-Study | Active Treatment Phase CC-90001 200mg Following Placebo PPF Sub-Study | Active Treatment Phase CC-90001 400mg Following Placebo PPF Sub-Study
All-Cause Mortality (participants affected / at risk) | 5/39 | 5/37 | 2/36 | 2/15 | 2/15 | 1/15 | 0/8 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 16/39 | 9/37 | 2/36 | 3/15 | 4/15 | 3/15 | 0/8 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 32/39 | 33/37 | 31/36 | 10/15 | 13/15 | 12/15 | 1/8 | 2/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CC-90001 200mg IPF Study (N=39) | CC-90001 400mg IPF Study (N=37) | Placebo IPF Study (N=36) | Active Treatment Phase CC-90001 200mg Following Placebo IPF Study (N=15) | Active Treatment Phase CC-90001 400mg Following Placebo IPF Study (N=15) | CC-90001 400mg PPF Sub-Study (N=15) | Placebo PPF Sub-Study (N=8) | Active Treatment Phase CC-90001 200mg Following Placebo PPF Sub-Study (N=3) | Active Treatment Phase CC-90001 400mg Following Placebo PPF Sub-Study (N=3)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Obstructive pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemophilus infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suspected COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CC-90001 200mg IPF Study (N=39) | CC-90001 400mg IPF Study (N=37) | Placebo IPF Study (N=36) | Active Treatment Phase CC-90001 200mg Following Placebo IPF Study (N=15) | Active Treatment Phase CC-90001 400mg Following Placebo IPF Study (N=15) | CC-90001 400mg PPF Sub-Study (N=15) | Placebo PPF Sub-Study (N=8) | Active Treatment Phase CC-90001 200mg Following Placebo PPF Sub-Study (N=3) | Active Treatment Phase CC-90001 400mg Following Placebo PPF Sub-Study (N=3)
Neutrophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 10 | 11 | 3 | 3 | 4 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 1 | 2 | 2 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 2 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 12 | 16 | 4 | 1 | 6 | 4 | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 6 | 7 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 3 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 3 | 0 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Herpes zoster (Infections and infestations) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 4 | 1 | 4 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 3 | 5 | 3 | 0 | 2 | 1 | 1 | 1 | 0
Post-acute COVID-19 syndrome (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Sialoadenitis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 5 | 4 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
Blood triglycerides increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Low density lipoprotein decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oxygen saturation decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 4 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 1 | 0 | 1 | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4 | 1 | 0 | 1 | 2 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 6 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 3 | 7 | 3 | 1 | 0 | 3 | 1 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 2 | 0 | 0 | 2 | 1 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Renal cyst (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 7 | 11 | 1 | 2 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 4 | 0 | 3 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 3 | 2 | 0 | 2 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0
Dependence on oxygen therapy (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Labyrinthitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urine cytology abnormal (Investigations) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypocholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ageusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT03142191/Prot_SAP_001.pdf